CLINICAL TRIAL: NCT04446195
Title: The Effect of Individualized Intervention on the Quality of Intestinal Preparation: a Randomized Controlled Study
Brief Title: The Effect of Individualized Intervention on the Quality of Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20200618
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Bowel Preparation Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group received routine intestinal preparation education.
- Experimental group (Active Comparator): The experimental group was treated with routine intestinal preparation education and individualized intervention.
  Interventions: Behavioral: Individualized Intervention

INTERVENTIONS:
Behavioral: Individualized Intervention — In this study, patients with the risk factors of insufficient intestinal preparation were treated with individualized intervention (mainly from the following aspects: chronic constipation, intestinal preparation not strictly in accordance with the requirements, body mass index > 25 kg / m2, age > 70 years old, with other diseases such as diabetes, Parkinson's disease, history of stroke or spinal cord injury, etc., application of tricyclic antidepressants or anesthetics).
  Arms: Experimental group

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignant tumors in the clinic. Colonoscopy is an important means of screening, diagnosis and treatment of colorectal diseases. The accuracy of diagnosis and the safety of treatment are closely related to the quality of intestinal preparation. Inadequate bowel preparation leads to poor effect of colonoscopy, which will reduce the effectiveness and safety of colonoscopy, increase the difficulty and time of colonoscopy, and increase the need of repeated colonoscopy. There are many factors that lead to poor bowel preparation. Recently, a number of studies at home and abroad have evaluated the risk factors related to insufficient bowel preparation. Obesity, men, older age, previous colon surgery history, accompanied by other diseases (such as diabetes, Parkinson's disease), taking antidepressants and other factors can affect the effect of bowel preparation. Although the research of intestinal preparation intervention and education methods has made a lot of progress, but in a series of reports, there are still a considerable number of patients in colonoscopy problems of intestinal preparation. At present, there are few researches on individualized intervention aiming at the risk factors of inadequate bowel preparation in China, so it is urgent to explore individualized bowel preparation scheme suitable for different populations. Therefore, the purpose of this experiment is to study individualized dryness aiming at the risk factors of insufficient bowel preparation in patients with the risk factors of insufficient bowel preparation The effect of pre-treatment on the quality of intestinal preparation can provide reference for improving the quality of intestinal preparation in patients with inadequate intestinal preparation.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a malignant tumor originates from colorectal mucosa epithelium. It is one of the most common malignant tumors in the world. Incidence rate of lung cancer is second only to lung cancer and breast cancer worldwide. In recent years, with the continuous improvement of people's living standard, changes in diet and diet structure and aging of population, the incidence rate and mortality rate of colorectal cancer in China have been increasing. A significant proportion of colorectal cancer patients have no characteristic clinical symptoms and reported symptoms. Many colorectal cancers have reached the middle and late stage when they are discovered, and their prognosis is poor. It can be seen that early prevention of colorectal cancer is very important. Timely screening for colorectal adenomas and endoscopic resection are the most effective measures to prevent colorectal cancer. Colonoscopy is currently recognized as the gold standard for colorectal cancer screening, which can not only detect early precancerous lesions, but also remove precancerous lesions and block the formation of colorectal cancer.Colonoscopy is an important means of screening, diagnosis and treatment of colonic diseases. The accuracy of diagnosis and the safety of treatment are closely related to the quality of intestinal preparation. Adequate intestinal preparation can make patients obtain higher intestinal cleanliness, ensure the integrity and correctness of colonoscopy, improve the detection rate of polyps and adenomas, increase the rate of cecal intubation and reduce the follow-up time The occurrence of adverse events such as shortened interval, intestinal perforation and missed diagnosis is of great significance for the realization of high-quality enteroscopy diagnosis and treatment.Bowel preparation is not a simple cathartic process, it involves all aspects of communication between patients and doctors. Good intestinal preparation includes following dietary restrictions before examination, applying adequate amount of appropriate cathartic drugs during intestinal preparation, waiting for the appropriate time interval between colonoscopies after intestinal preparation, and appropriate amount of active drinking water, etc. Strict dietary restriction and bowel cleaning are the necessary conditions to improve the quality of bowel preparation. Kang x et al. Showed that 18% to 30.5% of patients had insufficient bowel preparation [. Clinically, there may be more patients with poor bowel preparation. Inadequate bowel preparation will lead to longer operation time, more difficult catheterization of cecum, lower detection rate of adenoma and shorter follow-up time, which will increase the cost of colonoscopy. At present, Boston scale is widely used to evaluate the quality of intestinal preparation. The Boston scale divides the colon into three segments (cecum and ascending colon; hepatic, transverse and splenic flexure; descending, sigmoid and rectum). According to the worst-case to clean score, it is divided into four grades (0-3), with a total score of 0-9. Boston scale ≥ 6 points indicates that the intestinal preparation is qualified.There are many factors that lead to poor bowel preparation. Recently, a number of studies at home and abroad have evaluated the risk factors related to insufficient bowel preparation. Obesity, men, older age, previous colon surgery history, accompanied by other diseases (such as diabetes, Parkinson's disease), taking antidepressants and other factors can affect the effect of bowel preparation. Combined with the literature at home and abroad and the characteristics of Chinese people, the guidelines for gut preparation related to the diagnosis and treatment of digestive endoscopy in China suggest that the following factors are the risk factors for inadequate gut preparation in China: chronic constipation, failure to prepare the gut in strict accordance with the requirements (such as high fiber diet before operation, insufficient peg intake), body mass index > 25 kg / m2, age > 70 years old, colon surgery history With other diseases (such as diabetes, Parkinson's disease, history of stroke or spinal cord injury, etc.), application of tricyclic antidepressants or anesthetics.In addition, the guidelines for gut preparation related to the diagnosis and treatment of digestive endoscopy in China suggest that if the patient's gut preparation is not sufficient during the endoscopic examination, it should be actively evaluated and remedial measures should be taken or the endoscopic examination should be rescheduled. For the patients with the risk factors of insufficient intestinal preparation, other auxiliary measures can be taken to improve the intestinal preparation, such as the 4L peg program, low residue diet three days before endoscopic diagnosis and treatment, gastrointestinal motility promoting drugs, etc.; in addition, it is also of great value to further strengthen the education related to the optimization of intestinal preparation for the patients.In recent years, with the continuous development of China's economy, the continuous improvement of people's living conditions, and the continuous strengthening of patients' health awareness, colonoscopy has become one of the necessary items for many people's routine physical examination. However, in most medical institutions, when guiding patients to prepare for intestinal tract, there are some problems, such as lack of management, lack of detailed explanation, and complex process. These problems lead to the lack of understanding of intestinal tract preparation process for patients, thus affecting the preparation work before patients' examination and the follow-up treatment plan. Therefore, it has become one of the most important issues to study how to improve the intervention and guidance methods of patients' intestinal preparation and improve the quality of patients' intestinal preparation.Although the research of intestinal preparation intervention and education methods has made a lot of progress, various methods of intervention and guidance for patients before colonoscopy have been proposed at home and abroad to improve the quality of intestinal preparation. However, in a series of reports, there are still a considerable number of patients in the colonoscopy problems of intestinal preparation.At present, there are few researches on individualized intervention aiming at the risk factors of inadequate bowel preparation in China, so it is urgent to explore individualized bowel preparation programs suitable for different populations. Therefore, in this experiment, we designed individualized intervention for patients with insufficient bowel preparation (mainly from the following aspects: chronic constipation, not strictly in accordance with the requirements Bowel preparation, body mass index > 25 kg / m2, age > 70 years old, with other diseases such as diabetes, Parkinson's disease, history of stroke or spinal cord injury, application of tricyclic antidepressants or anesthetics). The purpose of the study is to study the effect of individualized intervention on the quality of intestinal preparation for patients with insufficient intestinal preparation, and to provide reference for improving the quality of intestinal preparation for patients with insufficient intestinal preparation.

ELIGIBILITY:
Inclusion criteria：

1. Aged between 18-75
2. Patients with insufficient bowel preparation
3. Patients without cognitive and communication barriers
4. Informed consent, voluntary participation in the study Exclusion criteria：

1. Severe suppurative inflammation of anus and rectum 2. Severe acute enteritis and ischemic enteropathy 3. After partial colorectal resection 4. Peritonitis, intestinal perforation, extensive adhesion in the abdominal cavity and intestinal stenosis caused by various reasons 5. Large abdominal aneurysm, highly abnormal bowel flexion and late cancer with extensive intraperitoneal metastasis 6. Dysphagia or impaired swallowing reflex 7. Obvious gastroparesis or gastric outlet obstruction or intestinal obstruction 8. Severe chronic renal failure (creatinine clearance < 30 ml / min) 9. Severe congestive heart failure (NYHA class III or IV) 10. Uncontrolled hypertension (systolic pressure > 170 mm Hg, diastolic pressure > 100 mm Hg) 11. Toxic colitis or megacolon 12. Disorder of water and electrolyte 13. Pregnancy or lactation 14. Mental patients 15. Failure to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation pass rate | During colonoscopy, endoscopists evaluated the quality of bowel preparation according to the Boston bowel preparation scale.
  The Boston Bowel preparation scale ≥6 indicates qualified intestinal preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Wang, MD, Principal Investigator — The Second Affiliated Hospital of Xi'an Jiaotong University,Xi'an, Shanxi, China
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China